CLINICAL TRIAL: NCT05182242
Title: Comparison of the Non-invasive Approach and Fetal Exome Sequencing in Prenatal Diagnosis When Fetal Ultrasound Signs Are Discovered
Acronym: DPNI-Exome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAMBOT PHRCI 2020
Record Dates: First submitted 2021-12-16; First posted 2022-01-10 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Antenatal Congenital Malformations
MeSH Terms: interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients (Experimental): Pregnant women with sonographic signs
  Interventions: Other: Collection of clinical data; Biological: Collection of samples; Other: Questionnaires; Other: Parent interviews
- Health professionals (Other): biologists, geneticists, obstetricians, midwives of the Pluridisciplinary Centers of Prenatal Diagnosis and genetic services
  Interventions: Other: Professional interview and focus groups

INTERVENTIONS:
Other: Collection of clinical data — family history, clinical data, ultrasound and all other data necessary for the study on a e-CRF (CleanWEB), allowing the collection of the family tree, and if necessary photographic elements.
  Arms: Patients
Biological: Collection of samples — Collected during fetal and blood sampling performed as part of care for ACPA:
  * 4 Streck tubes maximum for the pregnant woman for NIPD-Exome, collected prior to invasive fetal sampling
  * 1 additional vial of fetal sample (amniotic fluid or fetal blood) and 1 EDTA tube for each of the two parents
  Arms: Patients
Other: Questionnaires — within the framework of the pilot study (optional): questionnaires (about 20 minutes) for the evaluation of the experience, perceptions, impact of the analyses on the decision, satisfaction and concerns regarding exome sequencing (ES) and its results, opinion on certain types of results currently not reported, anxiety, possible psychological difficulties
  Arms: Patients
Other: Parent interviews — as part of the pilot study (optional): interview (about 1 hour) with a sociologist to explore perceptions of ES and the impact of the results, expectations about certain types of results that are not currently available, emotional situation, position regarding the continuation of the pregnancy
  Arms: Patients
Other: Professional interview and focus groups — Interview (approximately 45 minutes) to understand how the decision is formed Focus groups to help clarify whether the Variants of Unknown Significance (VUSs) should potentially be returned to the clinicians, or even the patient via the clinician
  Arms: Health professionals

SUMMARY:
The discovery of congenital malformations and/or non-specific signs by ultrasound (5% of pregnancies) represents a real medical challenge. Their prognosis is variable depending on the underlying etiology, ranging from acquired fetopathies to rare genetic diseases. In France, the diagnostic approach is currently based on imaging examinations (ultrasound, brain MRI, 3D bone scans, etc.) and/or biological examinations, generally on invasive sampling (trophoblast biopsy, amniocentesis or fetal blood puncture) with infectious (CMV, toxoplasmosis, parvovirus B19, etc.), metabolic (enzymes in the bloodstream, etc.), and genetic (standard karyotype, FISH, array CGH and targeted gene sequencing) investigations. The yield of this strategy is about 30%, leaving 70% of couples without a possible prognosis.

Over the last decade, medical genetics has undergone a technological revolution with the development of high-throughput DNA sequencing (HTS) allowing the analysis of targeted genes (panel) or the exome (ES). International studies published on the use of ES in prenatal diagnosis (PND) have become more common, with variable inclusion criteria, resulting in diagnostic rates between 15 and 36%, higher than those of array CGH (8-15%). In France, FHU TRANSLAD coordinates the national pilot study AnDDI-PRENATOME, which has made it possible to remove the technological barriers for PND ES and to obtain a diagnostic yield of 39% in 33 days on average.

In parallel, the recent development of NIPD (Non-invasive prenatal screening) on free fetal DNA circulating in maternal blood has made it possible to propose a non-invasive strategy. However, this technique is currently used in prenatal care only in a few indications: determination of the fetal sex, search for aneuploidies, analysis of the fetal rhesus status or, more rarely, the targeted diagnosis of monogenic diseases. The team in Strasbourg has recently conducted a pilot study using an NIPD-panel in couples with a history of neomutation in a gene responsible for intellectual disability, which has demonstrated the feasibility of capturing and then sequencing a panel of 500 genes on free fetal DNA circulating in maternal blood.

As high-depth exome sequencing from small amounts of DNA is now affordable and feasible, the investigators wish to compare invasive and non-invasive approaches for the discovery of fetal malformations on ultrasound: a trio exome analysis will be performed in parallel to circulating fetal DNA and fetal DNA extracted after an invasive puncture in order to compare the diagnostic performance of these two approaches.

The investigators propose a pilot study in order to prepare an organizational evaluation including an evaluation of the stakes for coordination and interactions between professionals, the relevance of the system (acceptability, expectations, satisfaction of couples and professionals...), its effectiveness and efficiency. The aim of this pilot project will be to observe the organizational impact on the Plurldisciplinary Centers for Prenatal Disagnostics and the genetic laboratories, and to refine the indicators necessary for monitoring the system; it will also involve conducting exploratory interviews with professionals and couples in order to prepare the qualitative study that will subsequently make it possible to evaluate the relevance of the organization.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with prenatal discovery of fetal malformations on ultrasound that may justify the performance of a fetal exome sequencing (e.g., multiple malformations and/or severe brain malformation, microphthalmia, bone damage, severe cardiac damage, etc.) who will have or are having an invasive prenatal sample for array CGA diagnosis and for which the results of the ES could change the outcome of the pregnancy
* Sufficient quantity of fetal sample (amniotic fluid or fetal blood or fetal DNA) for the collection of an additional sample for the ES
* Ability to collect blood samples from the pregnant woman and the biological father of the fetus (peripheral blood)
* Pregnant woman and father of the fetus aged ≥18 years
* Pregnant woman and father of the fetus able to comprehend the situation
* Person who has provided written consent

Exclusion Criteria:

* - Refusal of the pregnant woman or biological father to participate in the study
* Pregnancy before 11 weeks of amenorrhea or after 34 weeks of amenorrhea (to limit the risk of reporting results after birth)
* Pregnant women and/or biological fathers who are not affiliated to the national health insurance systel
* Pregnant women and/or biological fathers under some type of legal protection (guardianship, trusteeship, etc.)
* Pregnant women and/or biological fathers who are unable to express their consent

Organizational study:

In addition to the inclusion & exclusion criteria of the main study:

* Pregnant woman and/or biological father of fetus who provided oral consent to be interviewed
* Professionals (obstetrician, midwife, geneticist, biologist) willing to be interviewed or participate in a focus group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
number of etiological diagnosis common to the 2 analysis techniques : NIPD exomes and trio fetal ES | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Racine C, Garde A, Martz O, Safraou H, Eluard V, Rousseau T, Marle N, Harizay FT, Martin L, Maraval J, Bruel AL, Philippe C, Thauvin-Robinet C, Faivre L. First Prenatal Case of Genotypically and Phenotypically Overlapping Double Molecular Diagnosis of Van den Ende-Gupta and 22q11.2 Deletion Syndromes. Mol Genet Genomic Med. 2025 Apr;13(4):e70096. doi: 10.1002/mgg3.70096. PMID 40237608